CLINICAL TRIAL: NCT06424756
Title: Role of Mitochondria-derived Oxidative Stress on Microvascular Endothelial Function in Healthy Non-Hispanic Black and White Adults
Brief Title: Effects of an Antioxidant Supplement on Blood Vessel Health
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, S. Tony Wolf, Assistant Professor, University of Georgia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PROJECT00009286
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: Vascular dysfunction; Cardiovascular disease; Hypertension; Nitric oxide; Endothelial function
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension | interventions — mitoquinone; MitoTEMPO; tempol; NG-Nitroarginine Methyl Ester

STUDY DESIGN:
Intervention Model Description: For the experimental visits, participants will receive an antioxidant supplement in capsule form or a matching placebo pill in a randomized, double-blinded, crossover fashion. During each visit, participants will be given a single dose of the treatment to which they are randomized upon arrival at the laboratory (i.e., either 80 mg MitoQ or placebo will be administered on Visit 3, and the other treatment will be given on Visit 4). Peak concentrations of the antioxidant (MitoQ) occur after approximately 1 hour, allowing for appropriate time to prepare the participant for the experimental procedures.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MitoQ, then Placebo (Experimental): Participants will be given a single dose of 80mg MitoQ supplement first following an overnight fast. Then they will receive a matched Placebo single dose within a minimum 14 days
  Interventions: Dietary Supplement: MitoQ; Dietary Supplement: Placebo; Drug: MitoTempo; Drug: Tempol; Drug: L-NAME; Drug: SNP - Sodium Nitroprusside
- Placebo, then MitoQ (Experimental): Participants will be given a single dose of Placebo (matched to 80mg MitoQ) first following an overnight fast. Then they will receive 80mg MitoQ supplement single dose within a minimum of 14 days
  Interventions: Dietary Supplement: MitoQ; Dietary Supplement: Placebo; Drug: MitoTempo; Drug: Tempol; Drug: L-NAME; Drug: SNP - Sodium Nitroprusside

INTERVENTIONS:
Dietary Supplement: MitoQ — MitoQ supplement is composed of mitoquinol mesylate, which is a synthetic analog of coenzyme Q10
Dietary Supplement: Placebo — MitoQ matched Placebo
Drug: MitoTempo — During each experimental visit, intradermal microdialysis will be used to locally infuse MitoTempo (a mitochondria-specific superoxide dismutase mimetic) into the cutaneous microvasculature in the ventral aspect of the left forearm.
Drug: Tempol — During each experimental visit, intradermal microdialysis will be used to locally infuse Tempol (a superoxide dismutase mimetic) into the cutaneous microvasculature in the ventral aspect of the left forearm.
Drug: L-NAME — During each experimental visit, L-NAME (nitric oxide synthase inhibitor) will be perfused through microdialysis fibers for quantification of nitric oxide-mediated vasodilation.
Drug: SNP - Sodium Nitroprusside — At the end of each experimental visit, SNP will be perfused through microdialysis fibers to elicit a maximal vasodilation response.

SUMMARY:
Cardiovascular disease (CVD) is a leading cause of morbidity and mortality worldwide, and the non-Hispanic Black (NHB) population is disproportionately affected. Our research has previously demonstrated that oxidative stress may contribute to reduced vascular function in otherwise healthy NHB adults, potentially predisposing them to the development of hypertension and CVD. This study is designed to examine whether the mitochondria are an important source of oxidative stress-induced vascular dysfunction in healthy NHB adults.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as either non-Hispanic Black or non-Hispanic White.
* Men and women 18-75 years old.
* Non-hypertensive (systolic blood pressure [SBP]<130 and diastolic blood pressure [DBP] <85 mmHg).
* Have low density lipoprotein cholesterol <150mg/dl.
* Have HbA1C <6.0%.

Exclusion Criteria:

* Rash, skin disease, or disorders of pigmentation (e.g., psoriasis, eczema, vitiligo, or other skin inflammatory skin disorders)
* Known skin allergies to latex or adhesives
* Smoking and/or use of nicotine-containing products within the past year
* Use of illegal/recreational drugs
* Generalized kidney disease
* Taking chloramphenicol, cholestyramine, medication for seizures, methotrexate, nitrofurantoin, tetracycline, barbiturates, steroids, phenobarbital/phenytoin, orlistat or pyrimethamine
* Any current medications which could conceivably alter the cardiovascular control or responses
* Diagnosed or suspected metabolic or cardiovascular disease
* Current pregnancy or breastfeeding
* History of skin or other cancers
* Diagnosed or suspected diabetes (HbA1c ≥6.0)
* Anybody with narcolepsy or who has been diagnosed with any condition that impairs body temperature regulation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Cutaneous microvascular responses to local heating | 1 hour post intervention
  Using intradermal microdialysis, skin blood vessels will be locally treated with a mitochondria-targeted antioxidant (MitoTempo; 1 mM concentration). Nitric oxide (NO)-mediated skin vasodilation will be quantified via local inhibition of endothelial NO synthase during the course of the local skin heating protocol using L-NAME (15 mM concentration). Finally, maximal skin blood flow will be measured by heating the local area of skin to 43 degrees Celsius and locally perfusing sodium nitroprusside (SNP; an NO donor; 28 mM concentration). Two (2) thin fiber optic laser Doppler flowmeter probes and their holders, containing local heaters, will be used to measure skin blood flow.
Flow-mediated dilation responses | 1 hour post intervention
  FMD measures the health of blood vessels. The ultrasound makes sound waves to measure the size of blood vessels and the speed of the blood during rest and occlusion. The cuff is inflated to 220 mmHg (a commonly-used suprasystolic pressure; i.e., arterial blood flow is completely occluded) for 5 minutes to stop blood flow to and from the forearm.
Mitochondrial ROS production in peripheral blood mononuclear cells (PBMCs) | 1 hour post intervention
  Blood will be drawn for isolation of PBMCs and measurement of mitochondrial function and oxidative stress production.

CONTACTS AND LOCATIONS:
Locations (1):
- Ramsey Student Center, University of Georgia, Athens, Georgia, United States